CLINICAL TRIAL: NCT06925919
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety Tolerability and Pharmacokinetics of IDB-011 (IDB-774+IDB-898) in Healthy Adults
Brief Title: Study to Evaluate Safety, Tolerability and Pharmacokinetics of IDB-011
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: IDBiologics, Inc. (Industry)
Collaborators: Joint Program Executive Office Chemical, Biological, Radiological, and Nuclear Defense Enabling Biotechnologies (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IDB-RVFV-101
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Rift Valley Fever
Keywords: Healthy volunteer; Rift Valley fever virus
MeSH Terms: conditions — Rift Valley Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Experimental: IDB-011 Cohort 1 (Experimental): IDB-011 dose level 1
  Interventions: Drug: IDB-011 dose level 1
- Experimental: IDB-011 Cohort 2 (Experimental): IDB-011 dose level 2
  Interventions: Drug: IDB-011 dose level 2
- Experimental: IDB-011 Cohort 3 (Experimental): IDB-011 dose level 3
  Interventions: Drug: IDB-011 dose level 3
- Experimental: IDB-011 Cohort 4 (Experimental): IDB-011 dose level 4
  Interventions: Drug: IDB-011 dose level 4
- Experimental: IDB-011 Cohort 5 (Experimental): IDB-011 dose level 5
  Interventions: Drug: IDB-011 dose level 5
- Comparator: Placebo (Placebo Comparator): Normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IDB-011 dose level 1 — IDB-774 + IDB-898
  Arms: Experimental: IDB-011 Cohort 1
Drug: IDB-011 dose level 2 — IDB-774 + IDB-898
  Arms: Experimental: IDB-011 Cohort 2
Drug: IDB-011 dose level 3 — IDB-774 + IDB-898
  Arms: Experimental: IDB-011 Cohort 3
Drug: IDB-011 dose level 4 — IDB-774 + IDB-898
  Arms: Experimental: IDB-011 Cohort 4
Drug: IDB-011 dose level 5 — IDB-774 + IDB-898
  Arms: Experimental: IDB-011 Cohort 5
Other: Placebo — Normal saline
  Arms: Comparator: Placebo

SUMMARY:
Phase 1 randomized, double-blind, placebo-controlled trial to evaluate safety, tolerability, pharmacokinetics (PK) and immunogenicity of IDB-011 following intramuscular (IM )administration of single ascending doses to healthy adult participants.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo-controlled, dose escalation, first-in-human, Phase I clinical trial to assess the safety, tolerability, PK and immunogenicity of IDB-011 in healthy volunteers aged 18-64. IDB-011 is comprised of IDB-774 and IDB-898, which will be administered as separate, consecutive intramuscular injections.

Volunteers will be recruited into sequential dosing cohorts. Within each cohort, eligible volunteers will be randomly allocated (6:2) to receive either IDB-011 or placebo (0.9% normal saline). A sentinel dosing scheme will be employed for the first 2 volunteers in each dosing cohort.

Volunteers will stay in a clinical research unit for up to 4 consecutive days and be followed for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Body mass index (BMI) within 18.0 kg/m2 to 30.0 kg/m^2, inclusively
* Female participants must not be pregnant, breastfeeding or intend to become pregnant through 1 year post-administration
* Male subjects must agree to not cause pregnancy or donate sperm for 1 year post-administration
* Non-smoker
* Agree to abstain from alcohol for 72 hours and caffeine for 48 hours prior to administration and during the confinement period
* Agree to not donate blood or plasma during study participation
* Agree not to travel to Rift Valley fever virus (RVFV) endemic areas during participation

Exclusion Criteria:

* Known history of RVFV infection
* Previous receipt of RVFV vaccine
* Illness with fever within 5 days prior to administration
* History of malignancy within prior 5 years
* History of significant cardiovascular, pulmonary, gastrointestinal, liver, kidney, hematologic, neurological, psychiatric, endocrine, immunologic, dermatologic disease
* History of hypersensitivity reaction
* History or clinical evidence of alcohol abuse
* Human immunodeficiency virus (HIV) positive
* Hepatitis C virus positive
* Hepatitis B virus positive
* Received immunoglobulin or antibody product within 6 months of administration
* Vaccine within 28 days of administration
* Received investigational agent within 3 months or < 5 half-lives (whichever is longer) prior to administration
* Donation of plasma, 1 unit or > 500 mL blood donation in 56 days prior to administration

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability | Through 1 year from administration
  Safety to be measured via occurrence and severity of adverse events

SECONDARY OUTCOMES:
Characterize pharmacokinetic profile | Through 1 year from administration
  Concentration in serum over time
Evaluate immunogenicity | Through 1 year from administration
  Measurement of IDB-011 neutralizing antibodies in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Clinical Los Angeles, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No